CLINICAL TRIAL: NCT04094623
Title: The Muti-centered Investigation，Pathogenesis and Intervention Study of Non-suicidal Self-injury Behavior in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, Associate chief physician, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-KY043-01
Record Dates: First submitted 2019-09-04; First posted 2019-09-19 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: NSSI
MeSH Terms: interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSSI-DBT (Experimental): Dialectical behavior therapy, 2 hours every week for 13 weeks.
  Interventions: Other: Dialectical behavior therapy
- NSSI-SSGT (Active Comparator): Social support group therapy, 2 hours every week for 13 weeks.
  Interventions: Other: Social support group therapy

INTERVENTIONS:
Other: Dialectical behavior therapy — 15 patients in a group are treated by 2 psychotherapist by DBT including mindfulness skills, distress tolerance skills, emotional regulation skills and interpersonal effectiveness skills.
  Arms: NSSI-DBT
Other: Social support group therapy — 15 patients in a group are treated by 2 psychotherapist by SSGT.(Giving support to each other.)
  Arms: NSSI-SSGT

SUMMARY:
Non-suicidal self-injury (NSSINSSINSSI) refers to a series of direct and consequently repeated injuries to one's body without suicidal intent. At present, it has become an important issue of mental disorders. This study is expected to complete a multi-center epidemiological survey of non-suicidal self-injury in China, and to study its pathogenesis and intervention methods.

DETAILED DESCRIPTION:
(1) NSSI NSSI epidemiological survey. For example, epidemiological investigation. For example, in the period of 2020.1.1-2020.6.30 half a year, the psychiatric departments of fourteen hospitals of different regions, regions and nature (psychiatric specialist hospitals/general hospitals), hospitals of different types in Jiangsu Province, and hospitals of different types in Jiangsu Province were selected by stratification. In outpatient and inpatient departments, a certain proportion of young people were selected from outpatients and inpatients. Guided by the recommended diagnostic criteria of DSM-5 and guided by semi-structured interviews, the patients with NSSI behavior were screened out by semi-structured interviews. The incidence, comorbidity, incidence, comorbidity and basic psychosocial factors were investigated.(2) Exploring the pathogenesis of NSSI. Exploration of pathogenesis. A case-control study was designed on the basis of flow survey. The NSSI NSSI group and the normal control group were set up. The data of symptomatology, genetic factors of social factors of psychological cognitive function and brain imaging were collected. The data of brain imaging, brain imaging and other data were collected, and the data of social-psychological-biological data collection and mechanism exploration were carried out.(3) Clinical intervention study of NSSI. NSSI patients were randomly divided into structured DBT group intervention group (DBT-ST) and support group discussion group (SGT). The experimental group was given structured DBT group therapy intervention, while the control group was given the same frequency of support group discussion. To explore the therapeutic effect and mechanism of structured DBT group therapy intervention on NSSI behavior. In order to provide a scientific and effective treatment for NSSI behavior.

ELIGIBILITY:
Inclusion Criteria:

1. 10-40 years old;
2. Voluntary participation, signing informed consent and obtaining the consent of family members of patients under 18 years old;

Exclusion Criteria:

1. history and family of neurological or psychiatric disorders;
2. history of psychiatric disorders and family history;
3. severe somatic diseases;
4. taking psychotropic drugs within three months;
5. pregnancy and lactation

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-made Behavior Report Scale | 2 weeks
  Self reported non-suicidal self-injury behaviors over the past 2 weeks. Each item is scored 0-3(0=never; 3=every day), yielding a total between 0 and 6, also need choose locations of injury(such as hand, arm and so on. )

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lang AN, Zhong Y, Lei W, Xiao Y, Hang Y, Xie Y, Lv Z, Zhang Y, Liu X, Liang M, Zhang C, Zhang P, Yang H, Wu Y, Wang Q, Yang K, Long J, Liu Y, Wang S, Tang Y, Lei M, Zhang D, Ouyang L, Zhang L, Wang C. Neural mechanism of non-adaptive cognitive emotion regulation in patients with non-suicidal self-injury. Compr Psychiatry. 2024 Aug;133:152487. doi: 10.1016/j.comppsych.2024.152487. Epub 2024 May 1. PMID 38714144